CLINICAL TRIAL: NCT00229450
Title: Dose Response Effects of Estrogen Augmentation in Mood & Memory in Perimenopausal Depression
Brief Title: Estrogen and Perimenopausal Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NARSAD06806-001; 06806-001; 04-05-088
Record Dates: First submitted 2005-09-28; First posted 2005-09-29 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Depressive Disorder, Major; Menopause
Keywords: depression; menopause; perimenopause; mood; memory; perimenopausal; antidepressant; estrogen
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Estrogens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Treatment (Experimental): 0.625 mg/day of conjugated estrogen
  Interventions: Drug: Estrogen
- Placebo (Placebo Comparator): Daily placebo for conjugated estrogen
  Interventions: Drug: Estrogen

INTERVENTIONS:
Drug: Estrogen — 0.625 mg/day of conjugated Estrogen

SUMMARY:
During perimenopause (the time just prior to menopause), women often notice many biological, psychological, and social changes. In particular, some women experience depressive symptoms during perimenopause that are severe enough to warrant antidepressant medication. Whether or not women with perimenopausal depression respond to antidepressant medication may depend on the level of estrogen in their blood. This study will investigate whether estrogen will help women who only partially respond to antidepressant medications, as well as examine how different doses of estrogen may affect individuals differently.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Unipolar Major Depression, currently taking antidepressants
* HAM-D between 10 and 17

Exclusion Criteria:

* History of Psychosis, breast cancer, smoking, dementia, clotting disorders
* Current substance abuse

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2002-04; Primary Completion 2003-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Mood | 6 weeks
  17-item Hamilton Depression (HAM-D17) scores range from 0 to 50, and lower scores are better outcomes.

SECONDARY OUTCOMES:
Memory | 6 weeks
  The Buschke Selective Reminding Task (SRT) is a standardized measure of verbal learning that presents 12 words to the subject who is asked to immediately recall as many words as possible. The examiner then presents words that the subject was unable to recall until the subject can recall all 12 words without prompting twice, or until the examiner has presented prompts up to 12 times. Consistent Long-Term Retrieval score is the number of words that the subject recalls without receiving prompts and indicates how well the subject consolidates the new information during the learning phase (encoding). Scores indicate the sum of consistent long-term word retrieval across the 12 trials and range from 0 to 144, with higher scores indicating better learning.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda L. Morgan, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Neuropsychiatric Institute & Hospital, Los Angeles, California, United States

REFERENCES:
- [Background] Morgan ML, Cook IA, Rapkin AJ, Leuchter AF. Estrogen augmentation of antidepressants in perimenopausal depression: a pilot study. J Clin Psychiatry. 2005 Jun;66(6):774-80. doi: 10.4088/jcp.v66n0617. PMID 15960574
- [Background] Cook IA, Morgan ML, Dunkin JJ, David S, Witte E, Lufkin R, Abrams M, Rosenberg S, Leuchter AF. Estrogen replacement therapy is associated with less progression of subclinical structural brain disease in normal elderly women: a pilot study. Int J Geriatr Psychiatry. 2002 Jul;17(7):610-8. doi: 10.1002/gps.644. PMID 12112157